CLINICAL TRIAL: NCT06778343
Title: BIRDD: Biomarkers in Inflammatory Rheumatic Diseases Diagnosis - Ankylosing Spondylitis, Rheumatoid Arthritis and Systemic Lupus Erythematosus
Brief Title: Biomarkers in Inflammatory Rheumatic Diseases Diagnosis
Acronym: BIRDD
Status: Recruiting | Type: Observational
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Centro Hospitalar Lisboa Ocidental Hospital Egas Moniz (Unknown)
Responsible Party: Sponsor
Other Study IDs: CNTO1275ARA4001 (BIRDD)
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Ankylosing Spondylitis; Rheumatic Arthritis; Systemic Lupus Erythematosus
Keywords: Biomarker; Diagnosis
MeSH Terms: conditions — Spondylitis, Ankylosing; Rheumatic Fever; Lupus Erythematosus, Systemic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Peripheral Blood Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control
- Ankylosing Spondylitis
- Rheumatic Arthritis
- Systemic Lupus Erythematosus

SUMMARY:
Ankylosing spondylitis (AS), Rheumatoid Arthritis (RA) and Systemic Lupus Erythematosus (SLE) are three diseases where early diagnosis remains a major challenge. However, early diagnosis is the main determinant for a better prognosis. In the early stage, symptoms may be nonspecific and often difficult to establish a differential diagnosis between rheumatic diseases and other diseases, namely infectious and cancer diseases.

DETAILED DESCRIPTION:
The management of these diseases has undergone major advances in recent years, both in terms of the drugs armamentarium and therapeutic strategy. Treating disease to target, aiming at remission, through a tight control protocol is regarded as the standard of care. These principles were imported from RA and became the main strategy to approach several rheumatic inflammatory diseases. Reaching clinical and radiographic disease remission has therefore become an achievable goal. Increasing evidence has demonstrated that early diagnosis, prompt treatment initiation and early achievement of remission are the major predictors of good long-term clinical, functional and radiographic outcomes. The main reason for diagnostic delays is that classification criteria sets, including, imaging or biochemical changes, require time to occur. Rheumatoid factor, anti-CCP, ANA, anti-DNA and anti-Sm autoantibodies are often negative in the early stages of the disease; HLA B27 gene has a low specificity for AS. New criteria are now available and some biomarkers are emerging that allow earlier patient diagnosis. This new paradigm, needs new research trying to identify the most reliable biomarkers with relevance for clinical use.

The investigators intend to analyse biological samples, peripheral blood, from patients with well-established diagnosis (34 AS, 34 RA and 34 SLE) and 34 healthy controls (crossed by gender and age). Laboratory analysis will be based on transcriptomic approach trying to put in evidence specific biomarkers for each disease. The method is based on a analytical methodology already proven with success in stratifying patients.

The main objective of this study will be the development of a diagnostic chip to be implemented in clinical practice. The results should be confirmed in the same set of patients using quantitative real-time protein chain reaction (RT-PCR) and the validation in a new set of patients. The main objective of this project is to establish a quick method to stratify patients of the three diseases- AS, SLE, RA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AS, RA, SLE according the mentioned criteria;
* Ability to provide informed consent;
* If entering the study on NSAIDs, tramadol, combination of paracetamol and codeine or hydrocodone, and/or non-opioid analgesics, subject must be on stable dose(s) for at least 14 days prior to the screening visit;
* If entering the study on oral corticosteroids, subject must be on a stable dose of prednisone (≤ 10 mg/day), or oral corticosteroid equivalents, for at least 14 days prior to the screening visit;
* If entering the study on MTX, leflunomide, SSZ, and/or hydroxychloroquine, subject must be on a stable dose of MTX (≤ 25 mg/week) and/or SSZ (≤ 3 g/day) and/or hydroxychloroquine (≤ 400 mg/day) or leflunomide (≤ 20 mg/day) for at least 28 days prior to the screening visit. A combination of up to two background csDMARDs is allowed;
* Subject is judged to be in good health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, physical examination, x-Ray performed at the Screening Visit.

Exclusion Criteria:

* Current pregnancy or breastfeeding;
* Prior exposure to any biologic therapy;
* Intra-articular joint or tendon sheaths injections, spinal/paraspinal injection(s), or parenteral administration of corticosteroids within 28 days prior to the Baseline Visit. Inhaled or topical corticosteroids are allowed;
* Receipt of any live vaccine within 4 weeks prior to the screening visit;
* History of clinically significant (per Investigator's judgment) drug or alcohol abuse within the last 6 months;
* Subject has a history of inflammatory arthritis of different etiology other than AS, RA or SLE (including but not limited to PsA, mixed connective tissue disease, reactive arthritis, scleroderma, polymyositis, dermatomyositis, fibromyalgia), or any arthritis with onset prior to 17 years of age;
* Any uncontrolled medical condition (e.g., uncontrolled diabetes mellitus, unstable ischemic heart disease);
* History of any malignancy;
* Positive serology for hepatitis B, hepatitis C, or human immunodeficiency virus;
* Infections requiring hospitalization or intravenous treatment with antibiotics within 30 days or oral treatment with antibiotics within 14 days before enrollment;
* Note : Healthy Controls should be matched by gender and age. People with acute infections or injuries (in the last 6 months) or non-controlled chronic diseases (cardiac, metabolic, lung, neurologic, gastro-intestinal or renal) will be exclude. Family history of Auto-Immune diseases as diagnosed by a rheumatologist will be also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People that satisfy the eligibity criteria with AS, RA, SLE and healthy individuals (as controls) currently living in Portugal.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Identify a transcriptomic signature to optimize patient stratification (between AS, RA and SLE) | From enrollment to the end of the study at 12 weeks.

SECONDARY OUTCOMES:
Identify novel signaling pathways that may represent new therapeutic targets | From enrollment to the end of the study at 12 weeks.
Compare transcriptomic signatures in different levels of disease activity | From enrollment to the end of the study at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ULS Lisboa Ocidental, Hospital de Egas Moniz, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pimentel-Santos FM, Ligeiro D, Matos M, Mourao AF, Costa J, Santos H, Barcelos A, Godinho F, Pinto P, Cruz M, Fonseca JE, Guedes-Pinto H, Branco JC, Brown MA, Thomas GP. Whole blood transcriptional profiling in ankylosing spondylitis identifies novel candidate genes that might contribute to the inflammatory and tissue-destructive disease aspects. Arthritis Res Ther. 2011 Apr 7;13(2):R57. doi: 10.1186/ar3309. PMID 21470430
- [Result] Eilertsen GO, Becker-Merok A, Nossent JC. The influence of the 1997 updated classification criteria for systemic lupus erythematosus: epidemiology, disease presentation, and patient management. J Rheumatol. 2009 Mar;36(3):552-9. doi: 10.3899/jrheum.080574. Epub 2009 Jan 22. PMID 19208593
- [Result] van der Linden MP, Knevel R, Huizinga TW, van der Helm-van Mil AH. Classification of rheumatoid arthritis: comparison of the 1987 American College of Rheumatology criteria and the 2010 American College of Rheumatology/European League Against Rheumatism criteria. Arthritis Rheum. 2011 Jan;63(1):37-42. doi: 10.1002/art.30100. PMID 20967854
- [Result] van der Linden SM, Valkenburg HA, de Jongh BM, Cats A. The risk of developing ankylosing spondylitis in HLA-B27 positive individuals. A comparison of relatives of spondylitis patients with the general population. Arthritis Rheum. 1984 Mar;27(3):241-9. doi: 10.1002/art.1780270301. PMID 6608352
- [Result] Oglesby A, Korves C, Laliberte F, Dennis G, Rao S, Suthoff ED, Wei R, Duh MS. Impact of early versus late systemic lupus erythematosus diagnosis on clinical and economic outcomes. Appl Health Econ Health Policy. 2014 Apr;12(2):179-90. doi: 10.1007/s40258-014-0085-x. PMID 24573911
- [Result] Monti S, Montecucco C, Bugatti S, Caporali R. Rheumatoid arthritis treatment: the earlier the better to prevent joint damage. RMD Open. 2015 Aug 15;1(Suppl 1):e000057. doi: 10.1136/rmdopen-2015-000057. eCollection 2015. PMID 26557378
- [Result] Wendling D, Claudepierre P, Prati C. Early diagnosis and management are crucial in spondyloarthritis. Joint Bone Spine. 2013 Dec;80(6):582-5. doi: 10.1016/j.jbspin.2013.03.003. Epub 2013 Apr 8. PMID 23578940